CLINICAL TRIAL: NCT05202275
Title: The Optimization of Antiemetic Regimen for Chemoradiotherapy-induced Nausea and Vomiting (C-RINV) in Locally Advanced Head and Neck Squamous Cell Carcinoma (LA-HNSCCs): A Prospective Phase Ⅱ Trial
Brief Title: The Optimization of Antiemetic Regimen for C-RINV in LA-HNSCCs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ye Zhang, Clinical Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC2020A16
Record Dates: First submitted 2021-12-20; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Nausea; Vomiting; Head and Neck Squamous Cell Carcinoma; Radiotherapy Side Effect
Keywords: Chemoradiotherapy; nausea; vomiting; Antiemetic regimen
MeSH Terms: conditions — Nausea; Vomiting; Squamous Cell Carcinoma of Head and Neck; Radiation Injuries | interventions — Olanzapine; Palonosetron; Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OPA regimen (Experimental): All patients were given orally olanzapine 10mg once on d1-5; intravenously palonosetron 0.25mg once on d1; aprepitant 125 mg once on d1, then 80mg once on d2-5.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Intensity-modulated radiotherapy was given to the patients with regimen of 69.96 Gy-73.92 Gy to the gross target volume of nasopharynx, 69.96 Gy to the gross target volume of positive nodes, 60.06 Gy the high risk clinical target volume, 50.96 Gy to the low risk clinical target volume. Concurrent chemotherapy is administrated with cisplatin 100mg/m2 at d1, d22, d43 during radiotherapy. All patients were given orally olanzapine 10mg once on d1-5; intravenously palonosetron 0.25mg once on d1; aprepitant 125 mg once on d1, then 80mg once on d2-5 at every chemotherapy cycle.
  Other Names: Palonosetron; Aprepitant

SUMMARY:
This study sought to investigate the efficacy and safety of a three-drug combination antiemetic regimen of olanzapine combined with aprepitant and palonosetron for the prevention of chemoradiotherapy-induced nausea and vomiting in locally advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
Intensity modulated radiotherapy (IMRT) combined with high-dose cisplatin is the standard treatment for locally advanced head and neck squamous cell carcinoma. Previous clinical studies of concurrent chemoradiotherapy have shown that the incidence of nausea and vomiting after treatment with 5-HT3RA and dexamethasone is about 40%. Nausea and vomiting seriously affect the patient's treatment tolerance and quality of life. In our previous prospective phase 2 study (NCT03572829), the triple antiemetic regimen of NK-1R antagonist (aprepitant), dexamethasone and ondansetron was firstly used in patients with head and neck squamous cell carcinoma who received concurrent chemoradiotherapy. the primary endpoint-complete response rate was 86%, and the incidence of no vomiting was 88.4%, which was better than the data previously reported in the literatures. The incidence of no nausea was only 60.5%, and the hiccup caused by dexamethasone was as high as 16%. And with the confirmation of the efficacy of immunotherapy in head and neck squamous cell carcinoma, the use of dexamethasone may reduce immunotherapy. Therefore, it is necessary to further optimize the antiemetic regimen. In recent years, a number of randomized studies have confirmed that the addition of olanzapine can reduce the incidence of nausea and increase the complete response rate of high emetic chemotherapy. Other randomized studies have shown that in patients with malignant tumors (including head and neck squamous cell carcinoma and esophageal cancer) receiving concurrent chemoradiotherapy, the NK-1R antagonist was changed to olanzapine on the basis of the original triple regimen, which significantly redeced the incidence of nausea.

Therefore, on the basis of previous studies, this study intends to conduct a prospective, single-arm phase II study to explore the efficacy and safety of olanzapine combined with aprepitant and palonosetron in the prevention of nausea and vomiting in patients with locally advanced head and neck squamous cell carcinoma receiving IMRT and concurrent chemotherapy..

ELIGIBILITY:
Inclusion Criteria:

Pathology confirmed squamous cell carcinoma. The primary sites included nasopharynx, mouth, oropharynx, hypopharynx, larynx, nasal cavity and paranasal sinuses Aged 18 to 70 years old Stage III-IVB diseases Eastern Cooperative Oncology Group Performance Status 0-1 Normally functioning of liver, kidney, bone marrow Concurrent chemoradiotherapy is recommended after multi-disciplinary team discussion; Must be able to swallow tablets At least 12 weeks lifetime was expected; Fertile male or female patients volunteered to use effective contraception within 90 days of the study period and at the end of study.

Exclusion Criteria:

Other medical histories of malignancy apart from non-melanoma skin cancer, cervical carcinoma in situ, and early-stage cured prostate cancer Nausea and emesis occurred 24 hours before the start of CCRT Any medicine which affected metabolism through drug-metabolising enzymes CPY3A4 and CYP2D6 except for nighttime sedatives Mental and severe cognitive impairment Perinatal women or rejection of taking contraception during treatment Drug and/or alcohol addiction Symptomatic brain metastasis Gastrointestinal obstruction Hypocalcemia or any other conditions that could provoke emesis Treatment with another antipsychotic agent for 30 days before or during protocol therapy Concurrent chest or abdominal radiotherapy Concurrent use of corticosteroid or amifostine or quinolone antibiotic therapy Known hypersensitivity to olanzapine Known uncontrolled cardiac arrhythmia, uncontrolled congestive heart failure, or acute myocardial infarction within the previous 6 months Medical history of diabetic ketoacidosis or uncontrolled diabetes mellitus, prostate enlargement, narrow angle glaucoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Nausea-free response rate | Up to 6.5 weeks
  The percentage of patients with no nausea (Visual Analogue Scale score 0) during concurrent chemotherapy.

SECONDARY OUTCOMES:
Emesis-free response rate | Up to 6.5 weeks
  The percentage of patients with no emetic episodes during concurrent chemotherapy.
Complete response rate | Up to 6.5 weeks
  The percentage of patients with no emetic episodes and no use of rescue medication during concurrent chemotherapy.
Complete protection rate | Up to 6.5 weeks
  The percentage of patients with no emetic episodes, no use of rescue medication and significant nausea (Visual Analogue Scale score ≤25【0-100mm】)
The rate of no significant nausea | Up to 6.5 weeks
  The percentage of patients with no significant nausea (Visual Analogue Scale score ≤25【0-100mm】)

CONTACTS AND LOCATIONS:
Overall Officials: Ye Zhang, MD, Principal Investigator — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Ye Zhang, Beijing, Beijing Municipality, China